CLINICAL TRIAL: NCT02795286
Title: Automated Setting of Individualized Sodium Technology (ASIST) - Proof of Principle Study
Brief Title: Automated Setting of Individualized Sodium Technology
Acronym: ASIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1407-005
Record Dates: First submitted 2016-05-17; First posted 2016-06-10 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: End Stage Renal Disease (ESRD)
Keywords: Chronic Kidney Disease (CKD); End Stage Renal Disease (ESRD); Chronic Hemodialysis; In-center HD; Sodium; Isotonic Dialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- ASIST A (Experimental): Artis Haemodialysis Machine w/ ASIST Software - Isonatremic
  Interventions: Device: Artis Haemodialysis Machine w/ ASIST Software - Isonatremic
- ASIST B (Experimental): Artis Haemodialysis Machine w/ ASIST Software - Isotonic
  Interventions: Device: Artis Haemodialysis Machine w/ ASIST Software - Isotonic
- Conventional HD (Active Comparator): Artis Haemodialysis Machine w/o ASIST Software
  Interventions: Device: Artis Haemodialysis Machine w/o ASIST Software

INTERVENTIONS:
Device: Artis Haemodialysis Machine w/ ASIST Software - Isonatremic
  Arms: ASIST A
Device: Artis Haemodialysis Machine w/ ASIST Software - Isotonic
  Arms: ASIST B
Device: Artis Haemodialysis Machine w/o ASIST Software
  Arms: Conventional HD

SUMMARY:
The ASIST study is a medical device study testing the safety and efficacy of a new hemodialysis machine software in chronic haemodialysis patients. The software's intention is to reduce hemodialysis related symptoms such as unwell being, blood pressure changes by adapting the dialysis fluid ion concentration to the patients plasma ion concentration by conductivity measurement.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be in clinically stable condition as judged by the treating physician, and demonstrated by stable medical history, physical examination, and laboratory testing for 30 days prior to enrollment.
* Subject must be receiving HD or hemodiafiltration (HDF) for at least 30 days prior to study enrollment, be dialyzing a minimum of 3 times per week in an in-center setting and each treatment session must be between 3.5 and 5 hours in duration.
* Subject has a stable functioning vascular access (arteriovenous [AV] fistula, graft, or dual-lumen tunneled catheter) based on the judgment of the treating physician and is performing dual-needle therapy with an actual blood flow rate of 250 - 400 mL/min.
* Subject has a pre-dialysis plasma sodium of ≥132 mmol/L for at least 60 days prior to study enrollment.
* Subject has achieved a dialysis dose of stdKt/Vurea ≥ 2.1 within 60 days prior to enrollment.
* Subject has a pre-dialysis hemoglobin ≥ 90 g/L measured at Screening.

Exclusion Criteria:

* Female subjects who are pregnant, lactating, or planning to become pregnant during the study period.
* Subjects who have a significant psychiatric disorder or mental disability that could interfere with the subject's ability to provide Informed Consent and/or comply with protocol procedures.
* Subjects with a medical condition that the investigator thinks may interfere with the study objectives.
* Subjects with significant signs of access recirculation as judged by the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-03; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of Blood Pressure | Up to 9 weeks
Evaluation of Heart Rate | Up to 9 weeks
Occurrence of Hypotensive Episodes | Up to 9 weeks
Change in Plasma Sodium | Up to 9 weeks
Change in Plasma Tonicity | Up to 9 weeks
Change in MCV (Erythrocyte Mean Corpuscular Volume) | Up to 9 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Skane University Hospital, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No